CLINICAL TRIAL: NCT06526767
Title: Comparative Study of Different Dosages of Disposable Gastrointestinal Vibrating Capsule (Vibrabot Capsule) in the Treatment of Mild to Moderate Chronic Functional Constipation
Brief Title: Comparative Study of Different Dosages of Vibrabot Capsule in the Treatment of Chronic Functional Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, jiangxuan, Professor, Beijing Tsinghua Chang Gung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23648-4-01
Record Dates: First submitted 2024-07-14; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Chronic Functional Constipation
Keywords: Chronic Functional Constipation; Vibrating Capsule; Dose-response Relationship; Mechanism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Experimental): Subjects in control group took Vibrabot capsules twice a week, one pill/time (on Monday and Thursday), for six weeks.
  Interventions: Device: Vibrabot capsules twice a week
- Trial group 1 (Experimental): Subjects in trial group 1 took Vibrabot capsules three times a week, one pill/time (Monday, Wednesday, and Friday) for six consecutive weeks.
  Interventions: Device: Vibrabot capsules three times a week
- Trial group 2 (Experimental): Subjects in trial group 2 took Vibrabot capsules five times a week, one pill/time (Monday, Tuesday, Wednesday, Friday, and Saturday), for six weeks.
  Interventions: Device: Vibrabot capsules five times a week
- Trial group 3 (Experimental): Subjects in trial group 3 took Vibrabot capsules one pill/time, five times a week (Monday, Tuesday, Wednesday, Friday, and Saturday) during the first two weeks, three times a week (Monday, Wednesday, and Friday) during the middle two weeks, and two times a week (Monday and Thursday) during the last two weeks.
  Interventions: Device: Vibrabot capsules loading dose

INTERVENTIONS:
Device: Vibrabot capsules twice a week — Subjects in control group took Vibrabot capsules twice a week, one pill/time (on Monday and Thursday), for six weeks.
  Arms: Control group
Device: Vibrabot capsules three times a week — Subjects in trial group 1 took Vibrabot capsules three times a week, one pill/time (Monday, Wednesday, and Friday) for six consecutive weeks.
  Arms: Trial group 1
Device: Vibrabot capsules five times a week — Subjects in trial group 2 took Vibrabot capsules five times a week, one pill/time (Monday, Tuesday, Wednesday, Friday, and Saturday), for six weeks.
  Arms: Trial group 2
Device: Vibrabot capsules loading dose — Subjects in trial group 3 took Vibrabot capsules one pill/time, five times a week (Monday, Tuesday, Wednesday, Friday, and Saturday) during the first two weeks, three times a week (Monday, Wednesday, and Friday) during the middle two weeks, and two times a week (Monday and Thursday) during the last two weeks.
  Arms: Trial group 3

SUMMARY:
This is a single-center trial that enrolls 120 18- to 85-year-old patients with mild to moderate chronic functional constipation to study the dose-response relationship of the Vibrabot capsule as well as the mechanism of action of the Vibrabot capsule.

DETAILED DESCRIPTION:
This study was a single-center, prospective, randomized, parallel-controlled clinical trial. If a subject signs an Ethics Committee (EC)-approved study informed consent (ICF) that meets the inclusion criteria and does not meet any of the exclusion criteria, the subject is considered eligible for admission to the study. Participants with chronic functional constipation enrolled in the study completed a two-week baseline period in which they were advised to avoid taking any laxatives or other treatments for their constipation as much as possible. After the two-week basal period, all subjects were randomly assigned to the control group, trial group 1, trial group 2, and trial group 3 for the corresponding treatment.

Control group: Vibrabot capsule was taken twice a week, one pill/time (on Monday and Thursday), for six weeks; Trial group 1: Vibrabot capsule administration and dosage were three times a week, one pill/time (Monday, Wednesday, and Friday) for six consecutive weeks; Trial group 2: Vibrabot capsule administration and dosage five times a week, one pill/time (Monday, Tuesday, Wednesday, Friday, and Saturday), for six weeks; Trial group 3: Vibrabot capsule administration and dosage for the first two weeks, five times a week, one pill/time (Monday, Tuesday, Wednesday, Friday, and Saturday); for the middle two weeks, three times a week, one pill/time (Monday, Wednesday, and Friday); and for the last two weeks, two times a week, one pill/time (Monday and Thursday).

The subjects who receive Vibrabot capsules will undergo a neurotransmitter test and a fecal flora test before and after the treatment. After completion of treatment, subjects in each group entered a follow-up period, which was observed until the patient regained symptoms of constipation, i.e., when laxatives or other bowel-promoting treatments were used. If the subject never recovered from constipation, a minimum of 8 weeks of questionnaire completion was required, depending on the patient's compliance status. During the study period, the subjects are required to keep an e-diary recording daily bowel movements (BMs), medication intake, and discomforts, and complete the Patient Assessment of Constipation Symptoms (PAC-SYM) and the Patient Assessment of Constipation Quality of Life (PAC-QOL) questionnaires every two weeks. This study consists of a screening/baseline period, a treatment period, and a follow-up period. During the study, subjects are required not to change their diet and lifestyle.

Subjects are not expected to change their diet or lifestyle during the study. If the subject has not had a bowel movement for three or more consecutive days, the subject is allowed to use another method of defecation to assist with defecation. Subjects are required to avoid antibiotics, probiotics, prebiotics, and proton pump inhibitors throughout their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

- 1.18 to 85-year-old men and women. 2. People with moderate to severe functional constipation according to Rome IV criteria.

The Rome IV criteria for functional constipation are as follows:

1. Must include two or more of the following:

   * Straining during more than one-fourth (25%) of defecations;
   * Lumpy or hard stools (BSFS 1-2) more than one-fourth (25%) of defecations;
   * Sensation of incomplete evacuation more than one-fourth (25%) of defecations;
   * Sensation of anorectal obstruction/blockage more than one-fourth (25%) of defecations;
   * Manual maneuvers to facilitate more than one fourth (25%) of defecations (e.g., digital evacuation, support of the pelvic floor);
   * Fewer than 3 spontaneous bowel movements per week;
2. Loose stools are rarely present without the use of laxatives.
3. Insufficient criteria for irritable bowel syndrome Criteria fulfilled for the last three months with symptom onset at least six months prior to diagnosis.

Severity of constipation:

1. Mild: The symptoms are mild and do not affect daily life. Normal BMs can be restored through overall adjustment and medication use in a short time.
2. Moderate: The symptoms are between mild and severe symptoms.
3. Severe: The symptoms are severe and persistent, seriously affecting work and life, and requiring medications, and medications cannot be stopped, or medications are ineffective.

   3. People who had a colonoscopy within three years before screening and had negative results, or whose colonoscopy results are judged by the investigator as mild anomalies, but the cause of their constipation cannot be explained. If the colonoscopy report is unavailable, the study physician will determine if a colonoscopy is needed. If the subjects undergo a colonoscopy after signing the ICF, they will not enter the treatment period until their BMs return to the baseline level (which takes about 1-4 weeks).

   4. People had colonic polyps and a polypectomy (except for endoscopic submucosal dissection (ESD)). Those with a polyp ≤1 cm can be enrolled one month after the polypectomy. Those with a polyp >1 cm can be enrolled three months after the polypectomy.

   5. People who consent to participate in this trial, can communicate with the investigator, understand and comply with the relevant procedures and requirements during the study (including completing study questionnaires on time, being treated and visited as scheduled, and undergoing relevant examinations), and voluntarily sign the ICF.

   Exclusion Criteria:
   1. People who are not eligible for surgery or refuse to undergo any abdominal surgery.
   2. People with known or suspected gastrointestinal obstruction, stenosis, diverticulum, bleeding, malformation, and fistula.
   3. People allergic to polymeric materials.
   4. People implanted with cardiac pacemakers and using gastrointestinal pacemakers.
   5. People with abdominal aortic aneurysms, gastrointestinal vascular lesions, ulcers, and lesions with bleeding tendencies.
   6. People with dysphagia.
   7. People with severe depression and anxiety and severe acute gastrointestinal lesions.
   8. People who had gastrointestinal surgery or a history of surgery that changed the structure of the gastrointestinal tract (except for appendectomy) or people who underwent gastrointestinal ESD in the past three months.
   9. People with severe hemorrhoids (patients with grade III-IV hemorrhoids according to the Clinical Practice Guidelines for the Management of Hemorrhoids of the American Society of Colon and Rectal Surgeons).
   10. People who plan to undergo MRI in the near future.
   11. Pregnant women or women with pregnancy plans in the next year.
   12. People with other conditions, so the investigator considers them not eligible for this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportions of responders to the four therapies during the treatment period. | 6 weeks
  Responders are the subjects with an average increase of ≥1 complete spontaneous bowel movements (CSBMs) per week during the treatment period compared to the baseline period.

SECONDARY OUTCOMES:
The changes in neurotransmitter levels before and after treatment with Vibrabot capsules. | 6 weeks of treatment.
  Patients should have blood samples collected before and after treatment for the measurement of neurotransmitters such as Substance P (SP), Serotonin (5-HT), Nitric Oxide (NO), and Gamma-Aminobutyric Acid (GABA).
The changes in fecal microbiota before and after treatment with Vibrabot capsules. | 6 weeks of treatment.
  Patients should collect fecal specimens before and after treatment for the analysis of fecal microbiota species and abundance through 16S rRNA sequencing.
Assessment of quality of life among different treatment groups. | Every 2 weeks during the treatment period and the follow-up period, up to 14 weeks.
  The PAC-QOL questionnaire is the most validated tool for measuring the quality of life of patients with constipation. It consists of 28 self-reported items investigating the effects of constipation on the patient's quality of life in the past 2 weeks. The PAC-QOL questionnaire is subcategorized into 4 items on physical discomfort, 8 items on psychosocial discomfort, 5 items on treatment satisfaction, and finally 11 items on worries and discomfort. The response choice is on a Likert scale from 0 to 4. Higher scores mean higher negative effects on quality of life.
Assessment of the severity of patient-reported symptoms among different treatment groups. | Every 2 weeks during the treatment period and the follow-up period, up to 14 weeks.
  The PAC-SYM questionnaire has emerged as an important tool for assessing the severity of patient-reported symptoms of constipation. The 12-item questionnaire is divided into three symptom subscales: abdominal (four items); rectal (three items); and stool (five items). Items are scored on 5-point Likert scales, with scores ranging from 0 to 4 (0 ='symptom absent', 1 ='mild', 2 ='moderate', 3 ='severe', and 4 ='very severe'). A mean total score in the range of 0-4 is generated by dividing the total score by the number of questions completed; the lower the total score, the lower the symptom.
The proportions of responders to the four therapies during the follow-up period. | 8 weeks of follow-up.
  Responders are the subjects with an average increase of ≥1 complete spontaneous bowel movements (CSBMs) per week during the follow-up period compared to the baseline period.
The proportion of patients with complete spontaneous defecation (CSBM) ≥three times per week during the treatment period; | 6 weeks of treatment.
  Evaluating the proportion of patients with complete spontaneous defecation (CSBM) ≥three times per week among different treatment groups during the treatment period.
The proportion of patients with complete spontaneous defecation (CSBM) ≥three times per week during the follow-up period. | 8 weeks of follow-up.
  Evaluating the proportion of patients with complete spontaneous defecation (CSBM) ≥three times per week among different treatment groups during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Jiang, Professor, Principal Investigator — Beijing Tsinghua Changung Hospital
Locations (1):
- XuanJiang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No